CLINICAL TRIAL: NCT01205295
Title: Patient Anxiety and Concern as Predictors for the Perceived Quality and Efficacy of Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kolding Sygehus (Other)
Collaborators: Odense University Hospital (Other); University of Southern Denmark (Other)
Responsible Party: Ph.d. Stud. Randi Bilberg, Kolding Hospital
Other Study IDs: TBH-12-1106
Record Dates: First submitted 2010-09-13; First posted 2010-09-20 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2010-09

CONDITIONS: Anxiety; Orthopedic Surgery
Keywords: hip; shoulder; mental disorders; anxiety; concern; efficacy of treatment
MeSH Terms: conditions — Anxiety Disorders; Mental Disorders | interventions — Cognitive Behavioral Therapy; Papaverine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Mental disorders: Preoperative and postoperative screening of mental disorders and efficacy of treatment in hip and shoulder patient.
  Interventions: Other: Cognitive behavioural therapy

INTERVENTIONS:
Other: Cognitive behavioural therapy — Cognitive behavioural therapy Psychologist Preoperative Efficacy of treatment
  Other Names: Psychologist; Preoperative; Efficacy of treatment; Hip; Shoulder

SUMMARY:
Background: Previous studies have shown that anxiety and dissatisfaction with patient progress are predictors for increased postoperative pain and reduced impact and efficacy of pain treatment. However, it remains to be shown whether patient anxiety and concern are predictors for the perceived quality of patient progress and the perceived efficacy of treatment.

The aim of this study is to investigate whether there is a correlation between preoperative anxiety and concern, and the perceived quality and efficacy of postoperative treatment. The hypothesis is that anxious and concerned patients are less satisfied with treatment and have a poorer response of their treatment.

Methods/design: This PhD-project consists of four coherent studies. 1) A methodological study evaluating the CMD-SQ (Common Mental Disorder - Screening Questionnaire) questionnaire by a test-retest study. 2) The main study, a prospective follow-up study, has the aim of investigating the correlation between patient anxiety and concern, their perceived quality of patient progress and the perceived efficacy of treatment. This correlation will be detected by means of five questionnaires: CMD-SQ, EQ-5D, SF-12, HVOK, OHS or OSS. 3) A study consisting of an explicit internal medical audit with the aim to investigate whether the medical assessment of patient efficacy of treatment is consistent with their own self-reported efficacy of treatment. 4) An intervention study designed as a randomized clinical trial. The aim is to investigate whether a targeted effort towards patients with a high score of CMD-SQ, i.e. patients with anxiety and concern, can increase their self-reported efficacies of treatment and their perceived quality of progress. A total of 800 hip- and shoulder-patients will be included.

Discussion: If a correlation between patient anxiety and concern, their perceived quality of progress and the perceived efficacy of treatment is found, it will be relevant to screen all hip- and shoulder-patients for anxiety and concern preoperatively and deal with this before their operation. This study will provide a proposition of how these patients can be taken care of through cognitive behavioural therapy as a targeted effort towards their anxiety and concern.

Aim and hypothesis: The aim of this study is to investigate whether there is a correlation between patient anxiety and concern, and their perceived quality and efficacy of treatment. The overall hypothesis is that patients who are anxious and concerned are less satisfied with their treatment and have a poorer overall efficacy of their treatment.

ELIGIBILITY:
Inclusion Criteria:

* All hip- and shoulder-patients, who are referred for the first time to the Outpatient Department of Orthopaedic Surgery at Kolding Hospital, a part of Lillebaelt Hospital and Department of Orthopaedic Surgery, Odense University Hospital, Denmark are included.
* The patients must be able to speak and read Danish and must be at least 18 years old.
* To be included, they must enter a patient programme that implies an operation.

Exclusion Criteria:

* Patients with cancer or who are registered as terminal are excluded.
* Patients who have experienced a trauma within the past four weeks and those with a psychotic diagnosis are excluded, e.g. severe mental disorders such as schizophrenia, paranoid psychosis and bipolar affective disorders (DSM IV, F 20-29, F 30, 31).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hip and shoulder patients from the Department of Orthopaedic Surgery, Kolding Hospital, a part of Lillebaelt Hospital, Denmark and Department of Orthopaedics and Traumatology, Odense University Hospital, Denmark.
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2010-09; Primary Completion 2013-02 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Mental disorders. | Baseline(preoperative)
  CMD-SQ contains 38 items and was prepared as a tool for general practitioners to increase the focus on patient anxiety and concern. The questionnaire was translated into Danish and then validated without the test-retest. CMD-SQ consists of the following six subscales, each of them has been validated: SCL-AS, Whiteley-7, SCL-ANX4, SCL-8, SCL-DEF6 and CAGE. The patients respond on a Likert scale. A normal score is lower than four in the SCL-AS scale and no more than two in the remaining scales. A manual for assessing and validating the score of CMD-SQ is available.
Quality of life | Baseline (preoperative)
  EQ-5D is designed to assess the quality of life with no reference to a specific diagnosis. The questionnaire has been translated into Danish and validated. The scale includes five broad areas and a visual analogue scale. The self-reported health situation is reported on a scale from 0 to 100. The score 100 corresponds to the best self-reported health situation.
Self-reported health perception | Baseline (preoperative)
  SF-12 is an internationally and nationally validated questionnaire that evaluates patients' self-reported health perception. SF-12 is an abbreviated version of SF-36 and it contains 12 items, which are divided into physical and mental items. The patients respond on a Likert scale.
Function of the shoulder | Baseline (preoperative)
  The UK questionnaire Oxford Shoulder Score (OSS) are initially and similar, but related to two different categories of patients, namely shoulder - operated patients. The questionnaires are compiled in Oxford. Each questionnaire contains 12 items. The OSS has been translated into Danish and validated. The patients respond on a Likert scale from 1 - 5. The calculated scores can be between 12 and 60 points. 12 points reflects the best possible effect of treatment, and a score above 36 is categorized as an expression of a poor patient-assessed efficacy of treatment.
Function of the hip | Baseline (preoperative)
  The UK questionnaires Oxford Hip Score (OHS) are initially and similar, but related to two different categories of patients, namely THA operated patients. The questionnaires are compiled in Oxford. Each questionnaire contains 12 items. The OHS has been translated into Danish and is undergoing a validation process in a parallel project. The patients respond on a Likert scale from 1 - 5. The calculated scores can be between 12 and 60 points.

SECONDARY OUTCOMES:
Satisfaction with treatment | 3 day postoperative
  The Danish questionnaire HVOK deals with patients' priorities and satisfaction with treatment and is included in a revised form. Ten of the highest prioritised items were selected for this study. The patients respond on a Likert scale.
  The Royal College of Surgeons of England has developed the "Questionnaire for patients who have had hip surgery". The aim was to investigate patients´ satisfaction with surgery. It is relevant to select three items and use them as supplementary questions in this study. The patients respond on a Likert scale.
Mental disorders. | 3 months postoperative
  CMD-SQ contains 38 items and was prepared as a tool for general practitioners to increase the focus on patient anxiety and concern. The questionnaire was translated into Danish and then validated without the test-retest. CMD-SQ consists of the following six subscales, each of them has been validated: SCL-AS, Whiteley-7, SCL-ANX4, SCL-8, SCL-DEF6 and CAGE. The patients respond on a Likert scale. A normal score is lower than four in the SCL-AS scale and no more than two in the remaining scales. A manual for assessing and validating the score of CMD-SQ is available.
Quality of life | 3 months postoperative
  EQ-5D is designed to assess the quality of life with no reference to a specific diagnosis. The questionnaire has been translated into Danish and validated. The scale includes five broad areas and a visual analogue scale. The self-reported health situation is reported on a scale from 0 to 100. The score 100 corresponds to the best self-reported health situation.
Self-reported health perception | 3 months postoperative
  SF-12 is an internationally and nationally validated questionnaire that evaluates patients' self-reported health perception. SF-12 is an abbreviated version of SF-36 and it contains 12 items, which are divided into physical and mental items. The patients respond on a Likert scale.
Function of the shoulder | 3 months postoperative
  The UK questionnaire Oxford Shoulder Score (OSS) are initially and similar, but related to two different categories of patients, namely shoulder - operated patients. The questionnaires are compiled in Oxford. Each questionnaire contains 12 items. The OSS has been translated into Danish and validated. The patients respond on a Likert scale from 1 - 5. The calculated scores can be between 12 and 60 points. 12 points reflects the best possible effect of treatment, and a score above 36 is categorized as an expression of a poor patient-assessed efficacy of treatment.
Function of the hip | 3 months postoperative
  The UK questionnaires Oxford Hip Score (OHS) are initially and similar, but related to two different categories of patients, namely THA operated patients. The questionnaires are compiled in Oxford. Each questionnaire contains 12 items. The OHS has been translated into Danish and is undergoing a validation process in a parallel project. The patients respond on a Likert scale from 1 - 5. The calculated scores can be between 12 and 60 points.
Satisfaction with treatment | 3 months postoperative
  The Danish questionnaire HVOK deals with patients' priorities and satisfaction with treatment and is included in a revised form. Ten of the highest prioritised items were selected for this study. The patients respond on a Likert scale.
  The Royal College of Surgeons of England has developed the "Questionnaire for patients who have had hip surgery". The aim was to investigate patients´ satisfaction with surgery. It is relevant to select three items and use them as supplementary questions in this study. The patients respond on a Likert scale.
Mental disorders. | 12 months postoperative
  CMD-SQ contains 38 items and was prepared as a tool for general practitioners to increase the focus on patient anxiety and concern. The questionnaire was translated into Danish and then validated without the test-retest. CMD-SQ consists of the following six subscales, each of them has been validated: SCL-AS, Whiteley-7, SCL-ANX4, SCL-8, SCL-DEF6 and CAGE. The patients respond on a Likert scale. A normal score is lower than four in the SCL-AS scale and no more than two in the remaining scales. A manual for assessing and validating the score of CMD-SQ is available.
Quality of life | 12 months postoperative
  EQ-5D is designed to assess the quality of life with no reference to a specific diagnosis. The questionnaire has been translated into Danish and validated. The scale includes five broad areas and a visual analogue scale. The self-reported health situation is reported on a scale from 0 to 100. The score 100 corresponds to the best self-reported health situation.
Self-reported health perception | 12 months postoperative
  SF-12 is an internationally and nationally validated questionnaire that evaluates patients' self-reported health perception. SF-12 is an abbreviated version of SF-36 and it contains 12 items, which are divided into physical and mental items. The patients respond on a Likert scale.
Function of the shoulder | 12 months postoperative
  The UK questionnaire Oxford Shoulder Score (OSS) are initially and similar, but related to two different categories of patients, namely shoulder - operated patients. The questionnaires are compiled in Oxford. Each questionnaire contains 12 items. The OSS has been translated into Danish and validated. The patients respond on a Likert scale from 1 - 5. The calculated scores can be between 12 and 60 points. 12 points reflects the best possible effect of treatment, and a score above 36 is categorized as an expression of a poor patient-assessed efficacy of treatment.
Function of the hip | 12 months postoperative
  The UK questionnaires Oxford Hip Score (OHS) are initially and similar, but related to two different categories of patients, namely THA operated patients. The questionnaires are compiled in Oxford. Each questionnaire contains 12 items. The OHS has been translated into Danish and is undergoing a validation process in a parallel project. The patients respond on a Likert scale from 1 - 5. The calculated scores can be between 12 and 60 points.
Satisfaction with treatment | 12 months postoperative
  The Danish questionnaire HVOK deals with patients' priorities and satisfaction with treatment and is included in a revised form. Ten of the highest prioritised items were selected for this study. The patients respond on a Likert scale.
  The Royal College of Surgeons of England has developed the "Questionnaire for patients who have had hip surgery". The aim was to investigate patients´ satisfaction with surgery. It is relevant to select three items and use them as supplementary questions in this study. The patients respond on a Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Randi M Bilberg, Ph.d. stud., Study Chair — Kolding Sygehus
Locations (1):
- Department of Orthopaedics and Traumatology, Odense University Hospital, Odense, Odense, Denmark

REFERENCES:
- [Derived] Bilberg R, Norgaard B, Roessler KK, Overgaard S. Test-retest reliability of Common Mental Disorders Questionnaire (CMDQ) in patients with total hip replacement (THR). BMC Psychol. 2014 Sep 8;2(1):32. doi: 10.1186/s40359-014-0032-5. eCollection 2014. PMID 25685352
- [Derived] Bilberg R, Norgaard B, Overgaard S, Roessler KK. Patient anxiety and concern as predictors for the perceived quality of treatment and patient reported outcome (PRO) in orthopaedic surgery. BMC Health Serv Res. 2012 Aug 8;12:244. doi: 10.1186/1472-6963-12-244. PMID 22873940